CLINICAL TRIAL: NCT02444026
Title: Feasibility and Efficacy of an Internet-delivered Cognitive-behavioral Intervention for Insomnia in a National Cohort of Danish Breast Cancer Survivors
Brief Title: Feasibility and Efficacy of Internet-delivered CBT for Insomnia in a National Cohort of Danish Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2012-553-12
Record Dates: First submitted 2014-12-10; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2014-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iCBT for Insomnia (Experimental): The Internet intervention offered is the SHUT-i program (Sleep Healthy Using The Internet), which is based on the existing consensus concerning non-pharmacological treatment of insomnia and builds on previous validated CBT's for insomnia (CBT -I)
  Interventions: Behavioral: iCBT for Insomnia
- Control (No Intervention): The control group will be offered the intervention AFTER the study

INTERVENTIONS:
Behavioral: iCBT for Insomnia — Internet-delivered Cognitive Behavioural Therapy for Insomnia
  Arms: iCBT for Insomnia

SUMMARY:
The aim is, in a randomized controlled trial, to test the feasibility and evaluate the efficacy of an internet-based treatment for insomnia, previously tested in a group of 28 US cancer patients, in a large sample of Danish breast cancer survivors who are experiencing significant sleep problems 0-3 years after treatment. The investigators aim to test the following hypotheses: That a group receiving Internet-delivered cognitive-behavioral therapy (CCBT) for insomnia (CCBT-I) will experience reduced sleep latency, more hours of sleep, fewer awakenings during the night, improved sleep efficiency, increased subjective sleep quality, and improved quality of life after the intervention, when compared to a waiting list control group. The investigators also aim to explore a number of possible moderators of the effect (comorbidity, depression, fear of cancer recurrence tendency to ruminate) and mediating mechanisms (changes in sleep habits and sleep-related lifestyle factors).

DETAILED DESCRIPTION:
METHODS PARTICIPANTS

The participants are able, legally competent women, 18 years or older, from a national cohort of Danish women treated for primary breast cancer between 1st of June 2011 and 1st of Juli 2014:

Inclusion criteria: 1) Reported moderate-to-severe sleep disturbances, defined as a score> 5 on the Pittsburgh Sleep Quality Index (PSQI) (32;33) (see below), and 2) are found to be disease free. Furthermore, participants 3) are required to have access to the Internet.

Exclusion criteria: 1) Recurrence of breast cancer, 2) a second cancer, 3) and other serious physical or psychological comorbidity (e.g. depression, cardiovascular disease, and COPD), 4) shift work schedule, 5) other sleep disorders (sleep apnea, narcolepsy).

PROCEDURE INFORMATION AND REQUEST TO PARTICIPATE Women who fulfill the inclusion criteria and indicate an interest in receiving further information receive an information folder by post informing.

BASELINE MEASURES:

The baseline questionnaires contains questions about sleep quality, fatigue, depression, anxiety, quality of life, sleep habits and sleep-relevant lifestyles, together with use of health care services, sleep medication, and use of alternative medicine with the aim of treating sleep problems.

INTERVENTION:

The intervention program is designed to be completed in 6 weeks. To ensure that all participants have opportunity to complete the program they are granted access to the program for nine weeks .

POST-INTERVENTION:

After the intervention, participants in both groups are asked to complete a post-intervention questionnaire package and then to fill in the sleep diary for a 2-week period.

FOLLOW-UP:

After an additional 4 weeks both groups complete two sleep questionnaires (PSQI and the insomnia severity index) after which the waiting list group is offered the intervention.

INTERVENTION The Internet intervention offered is the SHUT-i program (Sleep Healthy Using The Internet), which is based on the existing consensus concerning non-pharmacological treatment of insomnia and builds on previous validated CBT's for insomnia (CBT -I) (34).

CONTROL GROUP Participants randomly assigned to the control condition are told that for practical reasons, they have to wait 15 weeks before partaking in the intervention.

PRIMARY ENDPOINTS A) Sleep diary (bedtime, sleep onset latency (SOL), number of awakenings, total length of awakenings, wake time, arising time, daytime naps, rating of soundness of previous night's sleep, rating of refreshed feeling upon morning awakening, and information about sleep aids : medication and/or alcohol use).

B) The Pittsburgh Sleep Quality Index (PSQI) (33). C) The Insomnia Severity Index (ISI) (39).

NUMBER OF PARTICIPANTS The combined effects found in the meta-analysis of published randomized trials of Internet-based treatment for insomnia (30) are: sleep quality (d=0.41), sleep efficiency (d=0.40), number of awakenings (d=-0.45), sleep onset latency (d=-0.55), total minutes slept (d=.22), time spent in bed (d=.25). If the investigators aim to detect an effect corresponding to an average of the effects above (d = 0.38) with 80% statistical power, at least 2 x 109 participants are required.

ETHICAL CONSIDERATIONS The investigators will adhere to the general ethical guidelines for human trials. All participants receive oral and written information about the project. They are informed that they can withdraw at any time from the study with no consequence for their current or future treatment. Participants are advised to continue any medical treatment for insomnia, and to consult a doctor before changing medical regimen.

PRIVACY AND DATA SECURITY The SHUT-I program stores any personal information in a separate one-way system that cannot be accessed from the Internet but only locally by the SHUT-i administrators. Connections between personal information and other data are encrypted. Data is stored physically on servers in locked facilities, in the United States.

ADVERSE EFFECTS, INCONVENIENCES, BENEFITS, AND RISKS The investigators do not expect Internet-based cognitive behavioral therapy to be associated with any adverse health effects or risks as no adverse effects has been reported for conventional CBT for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Reported moderate-to-severe sleep disturbances, defined as a score> 5 on the Pittsburgh Sleep Quality Index (PSQI).
* Disease free.
* Access to the Internet.

Exclusion Criteria:

* Recurrence of breast cancer
* A second cancer
* Other serious physical or psychological comorbidity (e.g. depression, cardiovascular disease, and COPD)
* Night work schedule
* Other sleep disorders (sleep apnea, narcolepsy) .

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Sleep diary | Up to 7 month
  The online sleep diaries contains 10 standard questions including information about bedtime, sleep onset latency (SOL), number of awakenings, total length of awakenings, wake time, arising time, daytime naps, rating of soundness of previous night's sleep, rating of refreshed feeling upon morning awakening, and information about sleep aids (medication and/or alcohol use).
The Pittsburgh Sleep Quality Index | Up to 7 month
The Insomnia Severity Index | Up to 7 month

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy (FACIT) | Up to 7 month
Beck's Depression Inventory (BDI-II) | Up to 7 month
State-Trait Anxiety Inventory (STAI) | Up to 7 month
EQ-5D | Up to 7 month
SF-12 | Up to 7 month
  Quality of life (QoL) is measured with the SF-12
Cognitive Failures Questionnaire (CFQ) | Up to 7 month
Sleep habits and sleep-relevant lifestyle | Up to 7 month
  Is assessed by adapting, further developing, and testing in the first phase of the study an existing instrument (Suzuki E, Tsuchiya M, Hirokawa K, Taniguchi T, Mitsuhashi T, Kawakami N. Evaluation of an internet-based self-help program for better quality of sleep among Japanese workers: a randomized controlled trial. J Occup Health 2008;50(5):387-99.), that measures: activities before bedtime, eating habits before bedtime, use of stimulants (coffee, tea, cola), alcohol, activities in the bedroom, exercise, thought patterns concerning sleep, etc.
Use of health services, self-help methods, sleep medication,fatigue, morningness-eveningness type, and complementary and alternative medicine/treatment | Up to 7 month
Pain (questionnaire) | Up to 7 month
  A short questionnaire assessing pain is included

OTHER OUTCOMES:
Moderator - Fear of Cancer Recurrence (FCR) | Up to 7 month
Moderator - Depressive symptoms (BDI-II) | Up to 7 month
Moderator - Charlson comorbidity index | Up to 7 month
Moderator -Emotional Control Scale (ECQ-R) | Up to 7 month
Moderator - The expected effects of and motivation to complete the intervention | Up to 7 month
  A short questionnaire has been developed to assess the expected effects of and motivation to complete the intervention
Moderator - Use of health services, self-help methods, sleep medication, and complementary and alternative medicine/treatment | Up to 7 month
Moderator - Pain | Up to 7 month
  A short questionnaire assessing pain has been developed
Moderator - Subjective response to a specific traumatic event | Up to 7 month
  The impact of event scale-revised (Weiss, D.S. The Impact of Event Scale-Revised. In J.P. Wilson, & T.M. Keane (Eds.), Assessing psychological trauma and PTSD: A practitioner'shandbook (2nd ed., pp. 168-189).2004. New York: Guilford Press
  ) is included as a measure of subjective response to a specific traumatic event. This scale approximates the DSM-IV criteria for posttraumatic stress disorder. Subjective response to both breast cancer and one other self-chosen traumatic event is assessed. The delineation of the self-chosen traumatic event is based on the traumatic life event questionnaire (TLEQ)
Moderator - Traumatic Life Events Questionnaire (TLEQ) | Up to 7 month
Mediator - Changes in sleep habits and sleep-related lifestyle from baseline to post-intervention | Up to 7 month
Mediator - The experience of and satisfaction with the intervention | Up to 7 month
  Weiss, D.S. The Impact of Event Scale-Revised. In J.P. Wilson, & T.M. Keane (Eds.), Assessing psychological trauma and PTSD: A practitioner'shandbook (2nd ed., pp. 168-189).2004. New York: Guilford Press Weiss, D.S. The Impact of Event Scale-Revised. In J.P. Wilson, & T.M. Keane (Eds.), Assessing psychological trauma and PTSD: A practitioner'shandbook (2nd ed., pp. 168-189).2004. New York: Guilford Press Measured by the instrument developed in the first trials of the SHUTi intervention (Thorndike FP, Saylor DK, Bailey ET, Gonder-Frederick L, Morin CM, Ritterband LM. Develop- ment and Perceived Utility and Impact of an Internet Intervention for Insomnia. E J Appl Psychol 2008;4(2):32-42.
  )

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, MDSci, Study Director — Unit for Psychooncology and Health Psychology Dept. of Oncology, Aarhus University Hospital and Dept of Psychology and Behavioural Science, Aarhus University
Locations (1):
- Unit for Psychooncology and Health Psychology, Dept. of Oncology, Aarhus University Hospital and Dept of Psychology and Behavioural Science, Aarhus University, Aarhus, Denmark, Denmark

REFERENCES:
- [Background] American Psychiatric Asssociation. Diagnostic and Statistical Manual of Mental Disor ders. Washington, DC: American Psychiatric Association; 2000.
- [Background] Ohayon MM. Epidemiology of insomnia: what we know and what we still need to learn. Sleep Med Rev. 2002 Apr;6(2):97-111. doi: 10.1053/smrv.2002.0186. PMID 12531146
- [Background] Buysse DJ. Insomnia state of the science: an evolutionary, evidence-based assessment. Sleep. 2005 Sep;28(9):1045-6. No abstract available. PMID 16268371
- [Background] Roth T. Insomnia: definition, prevalence, etiology, and consequences. J Clin Sleep Med. 2007 Aug 15;3(5 Suppl):S7-10. No abstract available. PMID 17824495
- [Background] Fiorentino L, Ancoli-Israel S. Sleep dysfunction in patients with cancer. Curr Treat Options Neurol. 2007 Sep;9(5):337-46. PMID 17716597
- [Background] Savard J, Ivers H, Villa J, Caplette-Gingras A, Morin CM. Natural course of insomnia comorbid with cancer: an 18-month longitudinal study. J Clin Oncol. 2011 Sep 10;29(26):3580-6. doi: 10.1200/JCO.2010.33.2247. Epub 2011 Aug 8. PMID 21825267
- [Background] Price MA, Zachariae R, Butow PN, deFazio A, Chauhan D, Espie CA, Friedlander M, Webb PM; Australian Ovarian Cancer Study Group; Australian Ovarian Cancer Study - Quality of Life Study Investigators. Prevalence and predictors of insomnia in women with invasive ovarian cancer: anxiety a major factor. Eur J Cancer. 2009 Dec;45(18):3262-70. doi: 10.1016/j.ejca.2009.05.030. Epub 2009 Jun 18. PMID 19540748
- [Background] Colagiuri B, Christensen S, Jensen AB, Price MA, Butow PN, Zachariae R. Prevalence and predictors of sleep difficulty in a national cohort of women with primary breast cancer three to four months postsurgery. J Pain Symptom Manage. 2011 Nov;42(5):710-20. doi: 10.1016/j.jpainsymman.2011.02.012. Epub 2011 May 26. PMID 21620648
- [Background] Hall M, Baum A, Buysse DJ, Prigerson HG, Kupfer DJ, Reynolds CF 3rd. Sleep as a mediator of the stress-immune relationship. Psychosom Med. 1998 Jan-Feb;60(1):48-51. doi: 10.1097/00006842-199801000-00011. PMID 9492239
- [Background] Irwin M. Effects of sleep and sleep loss on immunity and cytokines. Brain Behav Immun. 2002 Oct;16(5):503-12. doi: 10.1016/s0889-1591(02)00003-x. PMID 12401464
- [Background] Baron KG, Reid KJ, Kern AS, Zee PC. Role of sleep timing in caloric intake and BMI. Obesity (Silver Spring). 2011 Jul;19(7):1374-81. doi: 10.1038/oby.2011.100. Epub 2011 Apr 28. PMID 21527892
- [Background] Hairston KG, Bryer-Ash M, Norris JM, Haffner S, Bowden DW, Wagenknecht LE. Sleep duration and five-year abdominal fat accumulation in a minority cohort: the IRAS family study. Sleep. 2010 Mar;33(3):289-95. doi: 10.1093/sleep/33.3.289. PMID 20337186
- [Background] Vgontzas AN, Bixler EO. Short sleep and obesity: are poor sleep, chronic stress, and unhealthy behaviors the link? Sleep. 2008 Sep;31(9):1203. No abstract available. PMID 18788643
- [Background] Cappuccio FP, D'Elia L, Strazzullo P, Miller MA. Sleep duration and all-cause mortality: a systematic review and meta-analysis of prospective studies. Sleep. 2010 May;33(5):585-92. doi: 10.1093/sleep/33.5.585. PMID 20469800
- [Background] Dew MA, Hoch CC, Buysse DJ, Monk TH, Begley AE, Houck PR, Hall M, Kupfer DJ, Reynolds CF 3rd. Healthy older adults' sleep predicts all-cause mortality at 4 to 19 years of follow-up. Psychosom Med. 2003 Jan-Feb;65(1):63-73. doi: 10.1097/01.psy.0000039756.23250.7c. PMID 12554816
- [Background] Sleep complaints: Whenever possible, avoid the use of sleeping pills. Prescrire Int. 2008 Oct;17(97):206-12. PMID 19536941
- [Background] Belleville G. Mortality hazard associated with anxiolytic and hypnotic drug use in the National Population Health Survey. Can J Psychiatry. 2010 Sep;55(9):558-67. doi: 10.1177/070674371005500904. PMID 20840803
- [Background] Moore TA, Berger AM, Dizona P. Sleep aid use during and following breast cancer adjuvant chemotherapy. Psychooncology. 2011 Mar;20(3):321-5. doi: 10.1002/pon.1756. PMID 20878849
- [Background] van Straten A, Cuijpers P. Self-help therapy for insomnia: a meta-analysis. Sleep Med Rev. 2009 Feb;13(1):61-71. doi: 10.1016/j.smrv.2008.04.006. Epub 2008 Oct 26. PMID 18952469
- [Background] de Niet G, Tiemens B, Lendemeijer B, Hutschemaekers G. Music-assisted relaxation to improve sleep quality: meta-analysis. J Adv Nurs. 2009 Jul;65(7):1356-64. doi: 10.1111/j.1365-2648.2009.04982.x. Epub 2009 Apr 28. PMID 19456998
- [Background] Irwin MR, Cole JC, Nicassio PM. Comparative meta-analysis of behavioral interventions for insomnia and their efficacy in middle-aged adults and in older adults 55+ years of age. Health Psychol. 2006 Jan;25(1):3-14. doi: 10.1037/0278-6133.25.1.3. PMID 16448292
- [Background] Smith MT, Perlis ML, Park A, Smith MS, Pennington J, Giles DE, Buysse DJ. Comparative meta-analysis of pharmacotherapy and behavior therapy for persistent insomnia. Am J Psychiatry. 2002 Jan;159(1):5-11. doi: 10.1176/appi.ajp.159.1.5. PMID 11772681
- [Background] Morin CM, Culbert JP, Schwartz SM. Nonpharmacological interventions for insomnia: a meta-analysis of treatment efficacy. Am J Psychiatry. 1994 Aug;151(8):1172-80. doi: 10.1176/ajp.151.8.1172. PMID 8037252
- [Background] Ritterband LM, Bailey ET, Thorndike FP, Lord HR, Farrell-Carnahan L, Baum LD. Psychooncology 2011 Apr 29.
- [Background] Ritterband LM, Thorndike FP, Gonder-Frederick LA, Magee JC, Bailey ET, Saylor DK, Morin CM. Efficacy of an Internet-based behavioral intervention for adults with insomnia. Arch Gen Psychiatry. 2009 Jul;66(7):692-8. doi: 10.1001/archgenpsychiatry.2009.66. PMID 19581560
- [Background] Vincent N, Lewycky S. Logging on for better sleep: RCT of the effectiveness of online treatment for insomnia. Sleep. 2009 Jun;32(6):807-15. doi: 10.1093/sleep/32.6.807. PMID 19544758
- [Background] Suzuki E, Tsuchiya M, Hirokawa K, Taniguchi T, Mitsuhashi T, Kawakami N. Evaluation of an internet-based self-help program for better quality of sleep among Japanese workers: a randomized controlled trial. J Occup Health. 2008;50(5):387-99. doi: 10.1539/joh.l7154. Epub 2008 Aug 19. PMID 18716392
- [Background] Strom L, Pettersson R, Andersson G. Internet-based treatment for insomnia: a controlled evaluation. J Consult Clin Psychol. 2004 Feb;72(1):113-20. doi: 10.1037/0022-006X.72.1.113. PMID 14756620
- [Background] Riley WT, Mihm P, Behar A, Morin CM. A computer device to deliver behavioral interventions for insomnia. Behav Sleep Med. 2010;8(1):2-15. doi: 10.1080/15402000903425314. PMID 20043245
- [Background] Cheng SK, Dizon J. Computerised cognitive behavioural therapy for insomnia: a systematic review and meta-analysis. Psychother Psychosom. 2012;81(4):206-16. doi: 10.1159/000335379. Epub 2012 May 11. PMID 22585048
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Background] Beck SL, Schwartz AL, Towsley G, Dudley W, Barsevick A. Psychometric evaluation of the Pittsburgh Sleep Quality Index in cancer patients. J Pain Symptom Manage. 2004 Feb;27(2):140-8. doi: 10.1016/j.jpainsymman.2003.12.002. PMID 15157038
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] NIH State-of-the-Science Conference Statement on manifestations and management of chronic insomnia in adults. NIH Consens State Sci Statements. 2005 Jun 13-15;22(2):1-30. PMID 17308547
- [Background] Thorndike FP, Saylor DK, Bailey ET, Gonder-Frederick L, Morin CM, Ritterband LM. Development and Perceived Utility and Impact of an Internet Intervention for Insomnia. E J Appl Psychol. 2008;4(2):32-42. doi: 10.7790/ejap.v4i2.133. PMID 20953264
- [Background] Buysse DJ, Ancoli-Israel S, Edinger JD, Lichstein KL, Morin CM. Recommendations for a standard research assessment of insomnia. Sleep. 2006 Sep;29(9):1155-73. doi: 10.1093/sleep/29.9.1155. PMID 17040003
- [Background] Backhaus J, Junghanns K, Broocks A, Riemann D, Hohagen F. Test-retest reliability and validity of the Pittsburgh Sleep Quality Index in primary insomnia. J Psychosom Res. 2002 Sep;53(3):737-40. doi: 10.1016/s0022-3999(02)00330-6. PMID 12217446
- [Background] Thomsen DK, Mehlsen MY, Christensen S, Zachariae Rt. Pers Individ Diff 2003;34:1293-301.
- [Background] Morin CM. Insomnia: psychological assessment and management. New York: Guilford Press; 1993.
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Thorndike FP, Ritterband LM, Saylor DK, Magee JC, Gonder-Frederick LA, Morin CM. Validation of the insomnia severity index as a web-based measure. Behav Sleep Med. 2011;9(4):216-23. doi: 10.1080/15402002.2011.606766. PMID 22003975
- [Background] Savard MH, Savard J, Simard S, Ivers H. Empirical validation of the Insomnia Severity Index in cancer patients. Psychooncology. 2005 Jun;14(6):429-41. doi: 10.1002/pon.860. PMID 15376284
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Beck AT, Steer RA, Brown GK. Manual: Beck Depression Inventory. 2 ed. San Antonio, TX: The Psychological Corporation. Hartcourt & Brace.; 1996.
- [Background] Christensen S, Zachariae R, Jensen AB, Vaeth M, Moller S, Ravnsbaek J, von der Maase H. Prevalence and risk of depressive symptoms 3-4 months post-surgery in a nationwide cohort study of Danish women treated for early stage breast-cancer. Breast Cancer Res Treat. 2009 Jan;113(2):339-55. doi: 10.1007/s10549-008-9920-9. Epub 2008 Feb 16. PMID 18278553
- [Background] Spielberger CD. Psychological Assessment Resources Odessa FA 1988 1988.
- [Background] Zachariae R, Melchiorsen H, Frobert O, Bjerring P, Bagger JP. Experimental pain and psychologic status of patients with chest pain with normal coronary arteries or ischemic heart disease. Am Heart J. 2001 Jul;142(1):63-71. doi: 10.1067/mhj.2001.115794. PMID 11431658
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Bjørner JB, Damsgaard MT, Watt T, Bech P, Rasmussen NK, Kristensen TS, et al. Copenhagen: Lif; 1997.
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Katz JN, Chang LC, Sangha O, Fossel AH, Bates DW. Can comorbidity be measured by questionnaire rather than medical record review? Med Care. 1996 Jan;34(1):73-84. doi: 10.1097/00005650-199601000-00006. PMID 8551813
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Roger D, Najarian B. Pers Indiv Diff 1989;10(8):845-53.
- [Background] Weiss, D.S. The Impact of Event Scale-Revised. In J.P. Wilson, & T.M. Keane (Eds.), Assessing psychological trauma and PTSD: A practitioner'shandbook (2nd ed., pp. 168-189).2004. New York: Guilford Press.
- [Background] Kubany ES, Haynes SN, Leisen MB, Owens JA, Kaplan AS, Watson SB, Burns K. Development and preliminary validation of a brief broad-spectrum measure of trauma exposure: the Traumatic Life Events Questionnaire. Psychol Assess. 2000 Jun;12(2):210-24. doi: 10.1037//1040-3590.12.2.210. PMID 10887767
- [Background] O'Connor M, Christensen S, Jensen AB, Moller S, Zachariae R. How traumatic is breast cancer? Post-traumatic stress symptoms (PTSS) and risk factors for severe PTSS at 3 and 15 months after surgery in a nationwide cohort of Danish women treated for primary breast cancer. Br J Cancer. 2011 Feb 1;104(3):419-26. doi: 10.1038/sj.bjc.6606073. Epub 2011 Jan 11. PMID 21224851
- [Background] Pedersen CG, Christensen S, Jensen AB, Zachariae R. Prevalence, socio-demographic and clinical predictors of post-diagnostic utilisation of different types of complementary and alternative medicine (CAM) in a nationwide cohort of Danish women treated for primary breast cancer. Eur J Cancer. 2009 Dec;45(18):3172-81. doi: 10.1016/j.ejca.2009.09.005. Epub 2009 Oct 5. PMID 19811905
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Kenny DA, Kashy DA, Bolger N. Data analysis in social psychology. In: Gilbert D, Fiske S,Lindzey G, editors. The handbook of social psychology. 4 ed. Boston,MA: McGraw-Hill; 1998. p. 233-65.
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Sobel ME. Asymptotic intervals for indirect effects in structural equation models. In: Leinhart S, editor. Sociological methodology.San Francisco: Jossey-Bass; 1982. p. 290-312.
- [Background] Muller D, Judd CM, Yzerbyt VY. When moderation is mediated and mediation is moderated. J Pers Soc Psychol. 2005 Dec;89(6):852-63. doi: 10.1037/0022-3514.89.6.852. PMID 16393020
- [Background] Danmarks Statistik (Statistics Denmark). Befolkningens brug af internet (Internet use in the Danish population). Copenhagen: Danmarks Statistik (Statistics Denmark); 2011.
- [Background] Jensen-Johansen M, Christensen S, Valdimarsdottir H, Zakowski S, Bovbjerg DH, Jensen AB, et al. Unpublished manuscript 2010.
- [Background] Uniform requirements for manuscripts submitted to biomedical journals. International Committee of Medical Journal Editors. Ann Intern Med. 1997 Jan 1;126(1):36-47. doi: 10.7326/0003-4819-126-1-199701010-00006. No abstract available. PMID 8992922
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811